CLINICAL TRIAL: NCT00867113
Title: A Phase II, Non-Randomized, Open-Label Multicenter Study of 5 Year Adjuvant Imatinib Mesylate (Gleevec®) in Patients at Significant Risk for Recurrence Following Complete Resection of Primary Gastrointestinal Stromal Tumor (GIST)
Brief Title: Five Year Adjuvant Imatinib Mesylate (Gleevec®) in Gastrointestinal Stromal Tumor (GIST)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571BUS282
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Results first posted 2018-03-14 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Gastrointestinal Stromal Tumor (GIST)
Keywords: Imatinib; Protein Kinase Inhibitors; Gastrointestinal Stromal Tumors; Digestive System Diseases; Digestive System Neoplasms; Gastrointestinal Diseases; Gastrointestinal Neoplasms; Adjuvant; PERSIST; PERSIS-5
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Digestive System Diseases; Digestive System Neoplasms; Gastrointestinal Diseases; Gastrointestinal Neoplasms | interventions — Imatinib Mesylate

ARMS (1):
- Imatinib (Experimental): All subjects received in tablet form imatinib (STI571) 400 mg once daily.
  Interventions: Drug: imatinib mesylate

INTERVENTIONS:
Drug: imatinib mesylate — imatinib mesylate was supplied in 100 and 400 mg tablets

SUMMARY:
This is a Phase II, non-randomized, open-label, multi-center study conducted in the USA. The purpose of this trial is to evaluate the use of long term adjuvant imatinib mesylate in patients at significant risk for recurrence following complete resection of primary GIST.

DETAILED DESCRIPTION:
This is a Phase II, non-randomized, open-label, multi-center study conducted in the USA. The primary endpoint is to evaluate the use of long term adjuvant imatinib mesylate in patients at significant risk for recurrence following complete resection of primary GIST. A total of 85 adult patients, 18 years of age and older will be enrolled.Participants will take 400 mg of imatinib mesylate daily by mouth for a total of 5 years. At the conclusion of the treatment period, patients will be followed for 2 years for survival, status of response and antineoplastic treatments and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older.
2. Patient must have had a histological diagnosis of primary GIST.
3. The tumor must expressed KIT (CD117) protein by immunohistochemistry performed by central pathology.
4. Patient must have been at significant risk of tumor recurrence as defined by either:

   * Primary GIST (any site): ≥ 2 cm and a mitotic rate of ≥ 5/50 HPF's
   * Non-gastric primary GIST: ≥ 5cm
5. Patient must have undergone complete gross resection of a primary GIST within 12 weeks prior to first dose of imatinib study drug. The inclusion of R1 resections will be reviewed on a case by case basis by the Study Management Committee.
6. Patient must had no evidence of metastatic GIST on either 1) a post-operative CT of the abdomen and pelvis with intravenous and oral contrast or 2) MRI of the abdomen and pelvis with intravenous contrast. CT or MRI must have been performed within 8 weeks prior to first dose of imatinib study drug.
7. Performance status 0 or 1 (ECOG)
8. Patient must had the following post-operative laboratory values confirmed within 14 days prior to first dose of imatinib study drug:

   * total bilirubin < 1.5 x ULN NOTE: Patients with elevated bilirubin secondary to Gilbert's disease are eligible to participate in the study.
   * ALT and AST < 2.5 x ULN
   * creatinine < 1.5 x ULN
   * ANC > 1.5 x 109/L
   * platelets > 100 x 109/L
9. If patient is a cancer survivor, ALL of the following criteria apply:

   * Patient had undergone potentially curative therapy for all prior malignancies.
   * No evidence of any prior malignancies for at least 3 years with no evidence of recurrence (except for effectively treated basal cell or squamous carcinoma of the skin, carcinoma in-situ of the cervix that has been effectively treated by surgery alone, or lobular carcinoma in-situ of the ipsilateral or contralateral breast treated by surgery alone).
   * Patient is deemed by their treating physician to be at low risk for recurrence from prior malignancies.
10. Female patients of childbearing potential must have had negative pregnancy test within 7 days before initiation of study drug dosing. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential. Female patients of reproductive potential must have jagreed to employ an effective barrier method of birth control throughout the study and for up to 7 days following discontinuation of study drug.
11. Written, voluntary informed consent.

Exclusion Criteria:

1. Patient has metastatic GIST to the peritoneum, liver, lymph node, or other sites or recurrent GIST.
2. Prior treatment for GIST with the exception of prior treatment with imatinib adjuvant lasting ≤ 8 weeks following gross surgical resection.
3. Patient has received any other investigational agents within 28 days of first day of study drug dosing.
4. Patient with Grade III/IV cardiac problems as defined by the New York Heart Association Criteria. (i.e., congestive heart failure, myocardial infarction within 6 months of study)
5. Patients with severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risk or compromise compliance with the protocol (i.e., uncontrolled diabetes, chronic renal disease, chronic liver disease, or active uncontrolled infection).
6. Patient has a known diagnosis of human immunodeficiency virus (HIV) infection.
7. Patient receiving concurrent treatment with warfarin (acceptable alternative: low-molecular weight heparin).
8. Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2009-07-22 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2016-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- United States (21):
  - University of California San Diego - Moores Cancer Center Moores UCSD Cancer Center (31), La Jolla, California
  - University of Colorado University of Colorado, Aurora, Colorado
  - Washington Hospital Center Department of Medical Oncology, Washington D.C., District of Columbia
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Longstreet Cancer Center, Gainesville, Georgia
  - Kootenai Medical Center Kootenai Cancer Cancer, Coeur d'Alene, Idaho
  - North Shore University Health System, Evanston, Illinois
  - Dana Farber Cancer Institute Dana-Farber, Boston, Massachusetts
  - Karmanos Cancer Institute Karmonos Cancer Instit. (40), Detroit, Michigan
  - Washington University School of Medicine Center for Advanced Medicine, St Louis, Missouri
  - Southern Nevada Cancer Research Foundation S. Nevada Cancer Res (2), Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Cancer Center Memorial Sloan Kettering (7), New York, New York
  - Duke University Medical Center Duke University Med Ctr (8), Durham, North Carolina
  - Oregon Health & Science University OHS University, Portland, Oregon
  - Penn State University / Milton S. Hershey Medical Center Penn Stat University, Hershey, Pennsylvania
  - Roger Williams Medical Center Medical Center, Providence, Rhode Island
  - Kingport Hematology Oncology, Kingsport, Tennessee
  - MD Anderson Cancer Center/University of Texas MD Anderson Cancer Center (4), Houston, Texas
  - South Texas Oncology and Hematology, PA South Texas Onc/Hem, San Antonio, Texas
  - Virginia Oncology Associates Viriginia Oncology Assoc., Norfolk, Virginia

REFERENCES:
- [Derived] Raut CP, Espat NJ, Maki RG, Araujo DM, Trent J, Williams TF, Purkayastha DD, DeMatteo RP. Efficacy and Tolerability of 5-Year Adjuvant Imatinib Treatment for Patients With Resected Intermediate- or High-Risk Primary Gastrointestinal Stromal Tumor: The PERSIST-5 Clinical Trial. JAMA Oncol. 2018 Dec 1;4(12):e184060. doi: 10.1001/jamaoncol.2018.4060. Epub 2018 Dec 13. PMID 30383140
- [Derived] Essat M, Cooper K. Imatinib as adjuvant therapy for gastrointestinal stromal tumors: a systematic review. Int J Cancer. 2011 May 1;128(9):2202-14. doi: 10.1002/ijc.25827. PMID 21387287
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com/webapp/etrials/searchTrial.do?t=i&trialID=747&keywords=CSTI571BUS282

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total of 113 subjects were screened and 91 were enrolled..
Period: Treatment Period
Arm/Group | Imatinib
Started | 91
Safety Set | 91
Full Analysis Set (FAS) | 91
Completed | 46
Not Completed | 45
Not completed — Adverse Event | 15
Not completed — Death | 2
Not completed — Withdrawal by Subject | 19
Not completed — Lost to Follow-up | 3
Not completed — Administrative problems | 1
Not completed — Disease progression/relapse | 1
Not completed — Protocol Violation | 4
Period: Post Treatment After Survival Follow-up
Arm/Group | Imatinib
Started | 68
Completed | 57
Not Completed | 11
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 5
Not completed — Administrative problems | 4

BASELINE CHARACTERISTICS:
Arm/Group | Imatinib
Number analyzed (Participants) | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (12.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 48
ECOG Status [Count of Participants; unit: Participants] — ECOG 0 = Fully active, able to carry on all pre-disease performance without restriction; ECOG 1 =Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; ECOG 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; ECOG 3 = Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; ECOG 4 = Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair; ECOG 5 = Dead.
  Participants
    ECOG = 0 | 59
    ECOG = 1 | 32
Primary lesion location [Number; unit: participant] — Primary lesion
  participant
    Gastric | 50
    Duodenum | 4
    Jejunum ileum | 21
    Rectum | 1
    Other | 15
    Abdomen | 1
    Abdominal; Proximal Jejunal | 1
    Exact Location In Small Bowel Not Identified | 1
    Gastric Serosa-Min Invasion Outer Musc Prop | 1
    Ileum And Cecum | 1
    Pelvis - Organ Of Origin Unknown | 1
    Recto Vaginal | 1
    Retroperitoneal Mass | 1
    Sigmoid Colon | 1
    Small Bowel | 6

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-free Survival up to 60 Months
Description: Recurrence-free survival assessment is based on the radiologic evidence and is defined as the time from the date of first dose of imatinib to the date of the first documented disease recurrence or death due to any cause (event).
Time Frame: Baseline up to 60 months
Measure: Number; unit: participants with an event
Arm/Group | Imatinib
Number analyzed (Participants) | 91
participants with an event
  Subject with an event | 9
  Event = disease recurrence | 7
  Event=death | 2
  Subjects censored | 82

2. Primary Outcome: Kaplan-Meier Estimates for Recurrence-free Survival up to 60 Months
Description: Recurrence-free survival (RFS) assessment is based on the radiologic evidence and is defined as the time from the date of first dose of imatinib to the date of the first documented disease recurrence or death due to any cause (event). RFS estimates were summarized using the Kaplan-Meier product-limit method (Kaplan 1958). Censoring rules for RFS with the earliest occurring rule used in the analysis: subjects without objective recurrence of disease who were alive at the time of their discontinuation from study were censored at the end of study date or end of treatment visit date if the subject refused to be followed post treatment and subjects recording antineoplastic therapy during the study were censored on the date of the therapy initiated
Time Frame: Baseline up to 60 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Imatinib
Number analyzed (Participants) | 91
percentage of patients
  12 months | 97.7 [91.1 to 99.4]
  18 months | 97.7 [91.1 to 99.4]
  24 months | 96.5 [89.6 to 98.9]
  36 months | 95.1 [87.5 to 98.2]
  48 months | 95.1 [87.5 to 98.2]
  60 months | 90.1 [80.0 to 95.2]

3. Secondary Outcome: Overall Survival (OS) at 60 Months
Description: Overall survival was defined as the time from the date of the first dose of study drug to the date of death. Subjects who were alive at the time of discontinuation/completion of the study were censored at the end of study date or end of treatment visit date if the subject refused to be followed post treatment. Full analysis set.
Time Frame: Baseline up to approximately 60 months
Measure: Number; unit: participants
Arm/Group | Imatinib
Number analyzed (Participants) | 91
participants
  subjects who died | 3
  subjects censored | 88

4. Secondary Outcome: Kaplan-Meier Estimates for Overall Survival (OS) up to 60 Months
Description: as for outcome 3
Time Frame: Baseline up to appoximately 60 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Imatinib
Number analyzed (Participants) | 91
percentage of participants
  12 months | 100.00 [100.00 to 100.00]
  18 months | 100.00 [100.00 to 100.00]
  24 months | 98.0 [86.4 to 99.7]
  36 months | 98.0 [86.4 to 99.7]
  48 months | 98.0 [86.4 to 99.7]
  60 months | 93.8 [82.0 to 98.0]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit up to approximately 7 years
Groups:
- Imatinib: Imatinib
Arm/Group | Imatinib
Serious Adverse Events (participants affected / at risk) | 28/91
Other Adverse Events (participants affected / at risk) | 91/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib (N=91)
ANAEMIA (Blood and lymphatic system disorders) | 4
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1
CARDIAC FAILURE (Cardiac disorders) | 1
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 1
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 1
ABDOMINAL ADHESIONS (Gastrointestinal disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 2
COLITIS (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 1
GASTRIC ULCER (Gastrointestinal disorders) | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 2
PANCREATITIS (Gastrointestinal disorders) | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1
RETCHING (Gastrointestinal disorders) | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3
SMALL INTESTINAL PERFORATION (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 2
CHEST PAIN (General disorders) | 1
MALAISE (General disorders) | 2
PAIN (General disorders) | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 1
HYPERSENSITIVITY (Immune system disorders) | 1
ABDOMINAL INFECTION (Infections and infestations) | 1
APPENDICITIS (Infections and infestations) | 1
APPENDICITIS PERFORATED (Infections and infestations) | 1
CELLULITIS (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 1
PERITONITIS (Infections and infestations) | 2
PNEUMONIA (Infections and infestations) | 4
SIALOADENITIS (Infections and infestations) | 1
FALL (Injury, poisoning and procedural complications) | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 2
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1
OVERDOSE (Injury, poisoning and procedural complications) | 1
HEPATIC ENZYME INCREASED (Investigations) | 1
LIPASE INCREASED (Investigations) | 1
WEIGHT DECREASED (Investigations) | 1
DESMOID TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
HAIR FOLLICLE TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2
RADICULOPATHY (Nervous system disorders) | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1
CONFUSIONAL STATE (Psychiatric disorders) | 1
DELIRIUM (Psychiatric disorders) | 1
DEPRESSION (Psychiatric disorders) | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1
RENAL MASS (Renal and urinary disorders) | 1
URETERIC STENOSIS (Renal and urinary disorders) | 1
ALVEOLITIS (Respiratory, thoracic and mediastinal disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1
HYPERTENSION (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib (N=91)
ANAEMIA (Blood and lymphatic system disorders) | 15
LEUKOPENIA (Blood and lymphatic system disorders) | 6
NEUTROPENIA (Blood and lymphatic system disorders) | 8
VERTIGO (Ear and labyrinth disorders) | 7
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 6
LACRIMATION INCREASED (Eye disorders) | 5
PERIORBITAL OEDEMA (Eye disorders) | 31
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 5
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 5
ABDOMINAL PAIN (Gastrointestinal disorders) | 22
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 6
CONSTIPATION (Gastrointestinal disorders) | 7
DIARRHOEA (Gastrointestinal disorders) | 57
DYSPEPSIA (Gastrointestinal disorders) | 14
FLATULENCE (Gastrointestinal disorders) | 12
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 5
NAUSEA (Gastrointestinal disorders) | 65
VOMITING (Gastrointestinal disorders) | 34
CHILLS (General disorders) | 7
FATIGUE (General disorders) | 45
OEDEMA (General disorders) | 7
OEDEMA PERIPHERAL (General disorders) | 18
PAIN (General disorders) | 7
PYREXIA (General disorders) | 9
TEMPERATURE INTOLERANCE (General disorders) | 6
SINUSITIS (Infections and infestations) | 8
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 10
URINARY TRACT INFECTION (Infections and infestations) | 8
CONTUSION (Injury, poisoning and procedural complications) | 5
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 7
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 10
BLOOD BILIRUBIN INCREASED (Investigations) | 5
BLOOD CREATININE INCREASED (Investigations) | 6
NEUTROPHIL COUNT DECREASED (Investigations) | 6
WEIGHT INCREASED (Investigations) | 9
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 5
DECREASED APPETITE (Metabolism and nutrition disorders) | 12
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 5
HYPOKALAEMIA (Metabolism and nutrition disorders) | 10
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 6
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 14
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 16
BACK PAIN (Musculoskeletal and connective tissue disorders) | 11
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 5
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 37
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 5
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 11
MYALGIA (Musculoskeletal and connective tissue disorders) | 8
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 13
DIZZINESS (Nervous system disorders) | 17
DYSGEUSIA (Nervous system disorders) | 6
HEADACHE (Nervous system disorders) | 20
NEUROPATHY PERIPHERAL (Nervous system disorders) | 8
PARAESTHESIA (Nervous system disorders) | 6
SCIATICA (Nervous system disorders) | 5
DEPRESSION (Psychiatric disorders) | 8
INSOMNIA (Psychiatric disorders) | 8
COUGH (Respiratory, thoracic and mediastinal disorders) | 11
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 11
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 6
ALOPECIA (Skin and subcutaneous tissue disorders) | 9
DRY SKIN (Skin and subcutaneous tissue disorders) | 6
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 7
RASH (Skin and subcutaneous tissue disorders) | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial